CLINICAL TRIAL: NCT06191926
Title: Diagnostic Performance of Shear Wave Dispersive Imaging to Differenciate Benign From Malignant Breast Lesions: Comparison With Shear Wave Elastography
Brief Title: Diagnostic Performance of Shear Wave Dispersive Imaging in Breast Lesions: Comparison With Shear Wave Elastography
Status: Completed | Type: Observational
Sponsor: Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Bo Kyoung Seo, Professor, Korea University Ansan Hospital
Other Study IDs: DispersionUS
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — Shear-wave elastography and shear-wave dispersion ultrasound to evaluate the diagnostic performance of solid breast lesions for the diagnosis of breast cancer

SUMMARY:
Human soft tissue such as breast tissue has viscoelasticity property. However, most ultrasound has only been measured for elasticity and viscosity has been neglected. Shear wave elastography (SWE) is a ultrasound technique that quantifies tissue elasticity. Shear wave dispersion (SWD) imaging is a newly developed ultrasound technique that evaluates the dispersion slope of shear waves, which is related to the viscosity of biological tissues. The goal of this retrospective study was to compare diagnostic performance between SWE and SWD to distinguish benign from malignant breast masses and to investigate additional role of SWD. Using histological diagnosis of breast lesions as a standard reference, quantitative indices of SWE and SWD were evaluated to diagnose breast cancer, and the diagnostic performance of SWE and SWD was compared.

DETAILED DESCRIPTION:
This retrospective study was approved by our institutional review board, which waved the requrement for informed consent. The investigators obtained quantitative parameters of SWE and SWD of solid breast lesions before biopsy. The investigators measured average tumor elasticity and tumor-to-fat elasticity ratio on SWE and average tumor dispersion and tumor-to-fat ratio and on SWD from each breast lesion. Diagnostic performance of SWE and SWD was compared using the area under the curve (AUC), sensitivity, specificity, and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* patients with histological results

Exclusion Criteria:

* patients without histological results

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should fulfill the following criteria as follows:(a) histologically confirmed breast lesions and (b) shear wave elastography and dispersion ultrasound performed before biopsy
Sampling Method: Probability Sample
Enrollment: 594 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Elastography and dispersion parameters to determine benign or malignant tumors | baseline, pre-biopsy
  The elastography and dispersion ultrasound parameter values correlated with histological results.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Kyoung Seo, MD, PhD, Principal Investigator — Korea University
Locations (1):
- Bo Kyoung Seo, Ansan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided